CLINICAL TRIAL: NCT03888872
Title: Effect of High Tone Power Therapy on Neurophysiological Measures and Function Outcome in Patients With Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Ahmed Magdy Alshimy, Assistant Lecturer in Neurological Physical Therapy, October 6 University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/002261
Record Dates: First submitted 2019-03-22; First posted 2019-03-25 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Diabetic Neuropathy Peripheral

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Group I (Study): will consist of 20 patients with diabetic neuropathy and will receive High tone power therapy in addition to selected physical therapy program (Wobble board training, AROM exercises for both UL & LL, gentle manual stretching exercises for both UL & LL and graduated gait training). for 10 sessions every other day, each session for 1.45 hours (60 minutes for HiTop and 45 minutes for selected physical therapy program).
  Interventions: Device: High tone power therapy; Other: Selected Physical Therapy Program
- Group II (Experimental): Group II (Control): will consist of 20 patients with diabetic neuropathy and will receive selected physical therapy program only same as group I. For 10 sessions every other day, each session for 45 minutes.
  Interventions: Other: Selected Physical Therapy Program

INTERVENTIONS:
Device: High tone power therapy — 1- High Tone Power Therapy (HiTop 191): (For group I). The high tone power therapy through using a device (HiTop 191; gbo Medizintechnik, Rimbach, Germany).
  The intensity of the electrical stimulation will be adjusted to a pleasant level that did not produce any pain or discomfort. Duration: 60 min (Each one electrode to both thighs to the knee, each one electrode to both thighs to the groin). Position: lying / setting, Number of sessions: 10, Frequency of sessions: 3 times per week.
  Arms: Group I
Other: Selected Physical Therapy Program — Selected physical therapy program: (For both groups).
  1. Wobble board training:
  2. Active range of motion exercises (AROM):
  3. Gentle manual stretching exercises for both UL & LL:
  4. Graduated gait training:

SUMMARY:
The purpose of the study is to investigate the effect of high tone power therapy on neurophysiological measures and function outcome in patients with diabetic neuropathy.

DETAILED DESCRIPTION:
Diabetes is a chronic, metabolic disease characterized by elevated levels of blood glucose (or blood sugar), which leads over time to serious damage to the heart, blood vessels, eyes, kidneys, and nerves. The most common is type 2 diabetes, usually in adults, which occurs when the body becomes resistant to insulin or doesn't make enough insulin.

Diabetic neuropathies (DNs) are nerve damaging disorders associated with diabetes mellitus. These conditions are thought to result from diabetic microvascular injury involving small blood vessels that supply nerves (vasa nervorum) in addition to macrovascular conditions that can culminate in diabetic neuropathy.

The most common characteristics of diabetic neuropathy (DN) are a distal, symmetrical, primarily sensory polyneuropathy affecting the feet and legs in a chronic, slowly progressive manner. The incidence and prevalence of DN associated with duration of diabetes affect up to 50% of diabetic patients. Although DN is known as the most common complications of diabetes. Diabetic neuropathy is estimated that 40% to 50% of people with diabetes will have DN within 10 years of diagnosis.

High tone power therapy (Hi Top) is the percutaneous electrical stimulation of skeletal muscles using alternative frequencies between 4.096 and 32.768 hertz to produce a muscle contraction and the treatment of diabetic neuropathy. The therapy frequency is scanned with a defined frequency. This method is called SimulFAM for Simultaneous Frequency Amplitude Modulation.

High tone power therapy (Hi Top) is a new quantum leap in the field of electro therapy. It is Electrotherapy with sinusoidal alternating currents. The high tone power therapy provides a therapy with medium frequency sine waves. The therapy is free of direct current (D.C.) components. The amplitude and the frequency are modulated simultaneously. The higher the frequency, the more energy can be introduced corresponding to the individual threshold curve of the patient's electrosensitivity.

A short-term intervention over 5 days with HiTop has the potential to immediately reduce pain with a significantly stronger analgesic effect than TENS. Particularly, the first period of intervention showed that HTEMS reduces pain to a greater extent than TENS. From a clinical point of view, HTEMS showed a promising result, especially when comparing with TENS or considering the short period of intervention time.

SIGNIFICANCE OF THE STUDY:

Diabetic neuropathy is the most common complication of diabetes. It affects the feet and legs first, followed by the hands and arms. Signs and symptoms of peripheral neuropathy are often worse at night, and include: numbness or reduced ability to feel pain or temperature changes, tingling or burning sensation, sharp pain or cramps, muscle weakness, loss of reflexes especially in the ankle and loss of balance and coordination.

Sensory nerve action potential amplitude and conduction velocity (CV) have been shown to be sensitive indicators of nerve degeneration in patients with diabetes and have been used to detect DN. Diabetic neuropathy is associated with low sensory nerve amplitude potential (SNAP) and CV.

Recently shown in a pilot study that high tone power therapy stimulation of the thigh causing isometric muscle contraction might be an effective treatment for painful diabetic neuropathy.

High tone power therapy can stimulate a large number of nerves in the thigh, might therefore lead to a spinal stimulation that in turn decreases excitability of small nerve fibers and lead to improve function of diabetic neuropathy.

So, the current study is designed to investigate the effect of high tone power therapy on neurophysiological measures and function outcome in patients with diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Forty type II referred diabetic neuropathy patients from both genders their ages will be ranged from 40-60 years old.
2. All patients with diabetic neuropathy > 10 years having diabetes (will be examined according to the general and specific neurological evaluation sheet for diabetic neuropathy).
3. All patients in the study should be ambulant independently.
4. All patients should be medically stable.
5. The body mass index (BMI) ranged from 20:30 Kg/m2.
6. All patients will approve and sign a consent form.

Exclusion Criteria:

1. Patients < 10 years having diabetes.
2. Patients with musculoskeletal deformities and disorders.
3. Patients with psychiatric disorders or seizures.
4. Patients with visual and auditory impairment or tremors influencing balance.
5. Patients with other neuromuscular disorders.
6. Patients with BMI more than 30 kg/m2.
7. Patients with foot deformities and ulcers.
8. Patients with cognitive impairment using mini-mental state examination (MMSE).
9. Patients with lower limb operations.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2020-06-14 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Measuring Nerve Conduction Velocity | Up to 30 days
  Neuro pack M1 EP/EMG measuring system MEB-9200/9300

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University, El-Sheikh Zayed City, Giza Governorate, Egypt